CLINICAL TRIAL: NCT03149900
Title: Exploratory Evaluation of Biomarkers Associated With Treatment Response to Cosentyx (Secukinumab) in Psoriasis Patients
Acronym: BIOMARKER
Status: Completed | Type: Observational
Sponsor: Diamant Thaci (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Diamant Thaci, Prof. Dr. med., University of Luebeck
Organization: University of Luebeck (Other)
Other Study IDs: CAIN457ADE02T
Record Dates: First submitted 2016-11-30; First posted 2017-05-11 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Secukinumab: Patients will be recruited in the Comprehensive Center for Inflammation Medicine. The study population will consist of 40 subjects (both male and female), aged 18 years and older, in whom treatment with Secukinumab is clinically indicated and according to the licensed product specifications. The study drug will be prescribed by a doctor who is independent of this study. Visit 1 will be carried out prior to the first injection of Secukinumab.
  All patients will receive a number and the data will be recorded in a pseudo-anonymised form. No blinding is necessary for investigators or patients (open study), as all patients receive the same treatment (marketed product).
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — See Arm Description
  Other Names: Cosentyx

SUMMARY:
To identify possible genetic associations of clinical response to anti-IL-17A (Secukinumab) treatment in psoriasis using a combined gene association study and gene expression analysis.

To investigate the influence of IL-17A on the cutaneous microbial flora and to analyse cutaneous antimicrobial peptide expression in the skin of patients with psoriasis prior to, and during, treatment with Secukinumab to determine the extent to which the microbial flora is associated with response to treatment, as determined by the PASI75, PASI90, PGA- and DLQI improvement.

DETAILED DESCRIPTION:
Psoriasis vulgaris is a chronic inflammatory skin disease which is characterized by raised, well-demarcated, erythematous plaques and affects approximately 2% of the Caucasian population.

Patients suffering from moderate-to-severe psoriasis may be treated with a variety of systemic agents and treatment modalities, including retinoids, phototherapy and/or immunomodulatory drugs, including methotrexate, ciclosporin and fumarates. Patients are regularly monitored to determine the efficacy of treatment and to detect signs of systemic toxicity. Indeed, lack of efficacy and/or therapeutic toxicity are factors which require a re-evaluation of therapy. In addition to the conventional systemic treatments, systemic "biologic" therapies are playing an increasingly important role in the management of moderate to severe psoriasis.These treatments have resulted from advances in the understanding of the patho-physiology of psoriasis, combined with advances in molecular biology, in order to provide a more targeted therapy. Biologics include drugs targeting the production or signal transduction of tumour necrosis factor alpha (TNFα), and more recently, agents which target specific cytokines known to play an important role in the disease, including interleukin (IL) 12/23.

Despite these advances in psoriasis therapy, a relatively small number of patients initially fail to respond to biological psoriasis treatment or relapse during treatment. In fact, treatment with TNFα inhibitors and IL-12/23 monoclonal antibodies fails to induce disease control (PASI 75) in approximately 20-30% of the patients.

An alternative biological therapy, recently licensed for the management of moderate to severe psoriasis is Secukinumab (Cosentyx®). Secukinumab binds to human IL-17A and neutralizes the bioactivity of this cytokine. IL-17A is increasingly recognized as one of the principal pro-inflammatory cytokines in immune mediated inflammatory diseases, including psoriasis. A recombinant, high-affinity, fully human monoclonal anti-human IL-17A antibody of the IgG1/κ class, Secukinumab treatment has reportedly resulted in disease response rates of up to almost 80%, as measured by a 90% improvement in the Psoriasis Area and Severity Index measure (PASI). Moreover, treatment with Secukinumab was associated with superior improvements in quality of life indices (Dermatology Life Quality Index (DLQI) when compared to treatment with the IL12/23 inhibitor Ustekinumab. Given that treatment with biologics is reportedly associated with a loss of response over time, the development of novel classes of biologics, including those targeting IL-17, has been welcomed in terms of expanding the psoriasis treatment armamentarium.

Despite the clinical data supporting the use of Secukinumab in the management of moderate to severe psoriasis, there are currently no molecular tools to identify which patients are likely to respond to treatment. Identifying biomarker(s) of disease response would not only facilitate optimized and personalized treatment, but would also ensure that patients who are unlikely to respond are not exposed to the risks associated with biologic treatments, principally derived from long-term immunosuppression. In addition, given that psoriasis is often associated with several inflammatory diseases, including psoriatic arthritis and inflammatory bowel disease, such biomarkers may also serve a key role in predicting treatment response of those co-morbid conditions to biological therapy.

An interesting potential type of biomarker is the presence of single nucleotide polymorphisms (SNPs). Such polymorphisms are alterations in (i) genes which may be associated with genetic susceptibility to particular diseases or (ii) genes which are important in molecular pathways involved in disease and/or treatment response. Many respective genes in these pathways have been implicated by genome-wide association studies. For example, in terms of psoriasis, SNPs have been identified in cellular methotrexate efflux transporters which may influence both treatment response and the risk of methotrexate toxicity. On the other hand, variations in the genes important to the intracellular metabolism of methotrexate did not predict treatment response to methotrexate. Interestingly, variations in the IL17A and IL17A receptor gene are reportedly not associated with psoriatic arthritis susceptibility, although such variations remain to be systematically examined specifically in patients with psoriasis.

An additional potential type of biomarker is the cutaneous expression of anti-microbial peptides (AMPs). Initially identified in frog skin, AMP expression in human psoriatic skin, specifically human beta defensin 2, was identified almost two decades ago. Since then it has become clear that a range of AMPs are highly expressed in the involved skin of psoriatic patients compared to normal skin. These proteins serve a protective antimicrobial function in the skin, but at the same time they may also play an immunomodulatory role. Therefore, it is conceivable that they may influence the pathophysiology of psoriasis. Indeed, the AMP cathelicidin (LL37) was shown to modulate proinflammatory keratinocyte responses in vitro, leading the authors to speculate that LL37 "may promote IL17/IL22 and IL6 associated psoriasis.". Thus, it is at least possible that treatment with IL17-targetting biologics not only influences the cutaneous expression of AMPs, but also alters the cutaneous inflammatory milieu, which may in result in profound changes in the cutaneous bacterial flora which the skin supports.

To this end, a third promising type of biomarker is the presence and composition of the cutaneous bacterial flora; the skin microbiome. The term "cutaneous microbiome" describes the microbiological flora which colonizes human skin. There is evidence that the flora may be regulated in a time-, sex-, and medication-dependent manner. Indeed, describing and understanding the cutaneous microbiome is now the focus of intense research efforts to determine the role it may play in several skin diseases, including atopic dermatitis and bullous diseases.

Whilst several studies have suggested shifts in the microbiological composition in associated with psoriasis, relatively few studies have addressed longitudinal changes in the microbiome under therapy. Indeed, at present there are no studies which have specifically sought to identify changes in the cutaneous microbiome under IL17 targeted therapy. Given the importance of IL17 in the pathophysiology of psoriasis, this important gap in our knowledge needs to be urgently addressed.

Therefore, in summary, this study aims to identify and describe the presence of genetic variations governing susceptibility to psoriasis and response to treatment with secukinumab. This genetic data will be complemented by functional data determining gene expression before and during treatment and correlated with the expression of AMPs and the composition of the cutaneous microbiome. Using both genetic and phenotypic data we aim to identify novel biomarkers which can be rigorously tested and validated in subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give written, signed and dated informed consent before any study related activity is performed.
2. Chronic moderate to severe plaque type psoriasis for at least 6 months prior to baseline with a PASI score ≥ 10 and BSA ≥ 10 as per German guidelines.
3. Subjects must be at least 18 years of age at time of enrollment
4. Patients starting treatment with Secukinumab and for whom the clinical decision has been made prior to participation in the study.
5. Initiation of Secukinumab therapy, in patients who are not biologic naïve will be carried out according to a published consensus paper (Mrowietz et al. 2014)

Exclusion Criteria:

1. Exclusion criteria will comply with the licensed product specifications for Cosentyx (Secukinumab)
2. Patients incapable of giving full informed consent.
3. Forms of psoriasis other than chronic plaque-type at enrollment
4. Oral or topical antibiotic therapy within the month prior to enrollment
5. Phototherapy (UVB/PUVA) within the month prior to enrollment
6. Allergy to local anaesthetic or latex
7. Pregnancy/Lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 40 subjects (both male and female), aged 18 years and older, in whom treatment with Secukinumab is clinically indicated and according to the licensed product specifications. The study drug will be prescribed by a doctor who is independent of this study. Visit 1 will be carried out prior to the first injection of Secukinumab.
  All patients will receive a number and the data will be recorded in a pseudo-anonymised form. No blinding is necessary for investigators or patients (open study), as all patients receive the same treatment (marketed product).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Change in skin microbiome composition | from baseline to week 24
  Investigation of skin microbiome composition associated with treatment response in psoriasis patients treated with Secukinumab
Change in antimicrobial peptide composition | from baseline to week 24
  Investigation of antimicrobial peptide composition associated with treatment response in psoriasis patients treated with Secukinumab
Change in gene expression | from baseline to week 24
  Investigation of gene expression in RNA and DNA associated with treatment response in psoriasis patients treated with Secukinumab

CONTACTS AND LOCATIONS:
Overall Officials: Diamant Thaci, Prof. Dr., Principal Investigator — University of Luebeck
Locations (1):
- University Clinic Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schon MP, Boehncke WH. Psoriasis. N Engl J Med. 2005 May 5;352(18):1899-912. doi: 10.1056/NEJMra041320. No abstract available. PMID 15872205
- [Background] Johnson-Huang LM, Lowes MA, Krueger JG. Putting together the psoriasis puzzle: an update on developing targeted therapies. Dis Model Mech. 2012 Jul;5(4):423-33. doi: 10.1242/dmm.009092. PMID 22730473
- [Background] Langley RG, Elewski BE, Lebwohl M, Reich K, Griffiths CE, Papp K, Puig L, Nakagawa H, Spelman L, Sigurgeirsson B, Rivas E, Tsai TF, Wasel N, Tyring S, Salko T, Hampele I, Notter M, Karpov A, Helou S, Papavassilis C; ERASURE Study Group; FIXTURE Study Group. Secukinumab in plaque psoriasis--results of two phase 3 trials. N Engl J Med. 2014 Jul 24;371(4):326-38. doi: 10.1056/NEJMoa1314258. Epub 2014 Jul 9. PMID 25007392
- [Background] Tsoi LC, Spain SL, Knight J, Ellinghaus E, Stuart PE, Capon F, Ding J, Li Y, Tejasvi T, Gudjonsson JE, Kang HM, Allen MH, McManus R, Novelli G, Samuelsson L, Schalkwijk J, Stahle M, Burden AD, Smith CH, Cork MJ, Estivill X, Bowcock AM, Krueger GG, Weger W, Worthington J, Tazi-Ahnini R, Nestle FO, Hayday A, Hoffmann P, Winkelmann J, Wijmenga C, Langford C, Edkins S, Andrews R, Blackburn H, Strange A, Band G, Pearson RD, Vukcevic D, Spencer CC, Deloukas P, Mrowietz U, Schreiber S, Weidinger S, Koks S, Kingo K, Esko T, Metspalu A, Lim HW, Voorhees JJ, Weichenthal M, Wichmann HE, Chandran V, Rosen CF, Rahman P, Gladman DD, Griffiths CE, Reis A, Kere J; Collaborative Association Study of Psoriasis (CASP); Genetic Analysis of Psoriasis Consortium; Psoriasis Association Genetics Extension; Wellcome Trust Case Control Consortium 2; Nair RP, Franke A, Barker JN, Abecasis GR, Elder JT, Trembath RC. Identification of 15 new psoriasis susceptibility loci highlights the role of innate immunity. Nat Genet. 2012 Dec;44(12):1341-8. doi: 10.1038/ng.2467. Epub 2012 Nov 11. PMID 23143594
- [Background] Nair RP, Duffin KC, Helms C, Ding J, Stuart PE, Goldgar D, Gudjonsson JE, Li Y, Tejasvi T, Feng BJ, Ruether A, Schreiber S, Weichenthal M, Gladman D, Rahman P, Schrodi SJ, Prahalad S, Guthery SL, Fischer J, Liao W, Kwok PY, Menter A, Lathrop GM, Wise CA, Begovich AB, Voorhees JJ, Elder JT, Krueger GG, Bowcock AM, Abecasis GR; Collaborative Association Study of Psoriasis. Genome-wide scan reveals association of psoriasis with IL-23 and NF-kappaB pathways. Nat Genet. 2009 Feb;41(2):199-204. doi: 10.1038/ng.311. Epub 2009 Jan 25. PMID 19169254
- [Background] Gupta Y, Moller S, Zillikens D, Boehncke WH, Ibrahim SM, Ludwig RJ. Genetic control of psoriasis is relatively distinct from that of metabolic syndrome and coronary artery disease. Exp Dermatol. 2013 Aug;22(8):552-3. doi: 10.1111/exd.12192. PMID 23879815
- [Background] Rich P, Sigurgeirsson B, Thaci D, Ortonne JP, Paul C, Schopf RE, Morita A, Roseau K, Harfst E, Guettner A, Machacek M, Papavassilis C. Secukinumab induction and maintenance therapy in moderate-to-severe plaque psoriasis: a randomized, double-blind, placebo-controlled, phase II regimen-finding study. Br J Dermatol. 2013 Feb;168(2):402-11. doi: 10.1111/bjd.12112. PMID 23362969
- [Background] Thaci D, Blauvelt A, Reich K, Tsai TF, Vanaclocha F, Kingo K, Ziv M, Pinter A, Hugot S, You R, Milutinovic M. Secukinumab is superior to ustekinumab in clearing skin of subjects with moderate to severe plaque psoriasis: CLEAR, a randomized controlled trial. J Am Acad Dermatol. 2015 Sep;73(3):400-9. doi: 10.1016/j.jaad.2015.05.013. Epub 2015 Jun 17. PMID 26092291
- [Background] Batycka-Baran A, Maj J, Wolf R, Szepietowski JC. The new insight into the role of antimicrobial proteins-alarmins in the immunopathogenesis of psoriasis. J Immunol Res. 2014;2014:628289. doi: 10.1155/2014/628289. Epub 2014 May 8. PMID 24901012
- [Background] Chen YE, Tsao H. The skin microbiome: current perspectives and future challenges. J Am Acad Dermatol. 2013 Jul;69(1):143-55. doi: 10.1016/j.jaad.2013.01.016. Epub 2013 Mar 13. PMID 23489584
- [Background] Srinivas G, Moller S, Wang J, Kunzel S, Zillikens D, Baines JF, Ibrahim SM. Genome-wide mapping of gene-microbiota interactions in susceptibility to autoimmune skin blistering. Nat Commun. 2013;4:2462. doi: 10.1038/ncomms3462. PMID 24042968
- [Background] Glaser R, Harder J, Lange H, Bartels J, Christophers E, Schroder JM. Antimicrobial psoriasin (S100A7) protects human skin from Escherichia coli infection. Nat Immunol. 2005 Jan;6(1):57-64. doi: 10.1038/ni1142. Epub 2004 Nov 28. PMID 15568027
- [Background] Rothstein B, Gottlieb A. Secukinumab for treating plaque psoriasis. Expert Opin Biol Ther. 2016;16(1):119-28. doi: 10.1517/14712598.2016.1121986. Epub 2015 Dec 14. PMID 26577956
- [Background] Warren RB, Smith RL, Campalani E, Eyre S, Smith CH, Barker JN, Worthington J, Griffiths CE. Genetic variation in efflux transporters influences outcome to methotrexate therapy in patients with psoriasis. J Invest Dermatol. 2008 Aug;128(8):1925-9. doi: 10.1038/jid.2008.16. Epub 2008 Feb 7. PMID 18256692
- [Background] Warren RB, Smith RL, Campalani E, Eyre S, Smith CH, Barker JN, Worthington J, Griffiths CE. Outcomes of methotrexate therapy for psoriasis and relationship to genetic polymorphisms. Br J Dermatol. 2009 Feb;160(2):438-41. doi: 10.1111/j.1365-2133.2008.08898.x. Epub 2008 Oct 25. PMID 19016697
- [Background] Catanoso MG, Boiardi L, Macchioni P, Garagnani P, Sazzini M, De Fanti S, Farnetti E, Casali B, Chiarolanza I, Nicoli D, Luiselli D, Salvarani C. IL-23A, IL-23R, IL-17A and IL-17R polymorphisms in different psoriatic arthritis clinical manifestations in the northern Italian population. Rheumatol Int. 2013 May;33(5):1165-76. doi: 10.1007/s00296-012-2501-6. Epub 2012 Sep 7. PMID 22955875
- [Background] Harder J, Bartels J, Christophers E, Schroder JM. A peptide antibiotic from human skin. Nature. 1997 Jun 26;387(6636):861. doi: 10.1038/43088. No abstract available. PMID 9202117
- [Background] Chen X, Takai T, Xie Y, Niyonsaba F, Okumura K, Ogawa H. Human antimicrobial peptide LL-37 modulates proinflammatory responses induced by cytokine milieus and double-stranded RNA in human keratinocytes. Biochem Biophys Res Commun. 2013 Apr 19;433(4):532-7. doi: 10.1016/j.bbrc.2013.03.024. Epub 2013 Mar 20. PMID 23524263
- [Background] Alekseyenko AV, Perez-Perez GI, De Souza A, Strober B, Gao Z, Bihan M, Li K, Methe BA, Blaser MJ. Community differentiation of the cutaneous microbiota in psoriasis. Microbiome. 2013 Dec 23;1(1):31. doi: 10.1186/2049-2618-1-31. PMID 24451201
- [Background] Statnikov A, Alekseyenko AV, Li Z, Henaff M, Perez-Perez GI, Blaser MJ, Aliferis CF. Microbiomic signatures of psoriasis: feasibility and methodology comparison. Sci Rep. 2013;3:2620. doi: 10.1038/srep02620. PMID 24018484
- [Background] Mrowietz U, de Jong EM, Kragballe K, Langley R, Nast A, Puig L, Reich K, Schmitt J, Warren RB. A consensus report on appropriate treatment optimization and transitioning in the management of moderate-to-severe plaque psoriasis. J Eur Acad Dermatol Venereol. 2014 Apr;28(4):438-53. doi: 10.1111/jdv.12118. Epub 2013 Feb 26. PMID 23437792